CLINICAL TRIAL: NCT01019694
Title: Patient Acceptability of Ipratropium Bromide/Albuteroll Delivered by the Respimat® Inhaler in Adults With Chronic Obstructive Pulmonary Disease
Brief Title: Combivent Respimat 1-year Safety Study in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1012.62
Record Dates: First submitted 2009-11-16; First posted 2009-11-25 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol, Ipratropium Drug Combination; Ipratropium

ARMS (3):
- Combivent Respimat 20/100 microgram(mcg) (Experimental): patient to take 1 inhalation 4 times a day
  Interventions: Drug: Combivent Respimat 20/100 mcg
- Combivent CFC-MDI 36/206 microgram-mcg (Active Comparator): patient to take 2 inhalations 4 times a day
  Interventions: Drug: Combivent CFC-MDI
- Atrovent HFA 42 mcg + Albuterol HFA (Active Comparator): patient to take 2 inhalations of each 4 times a day
  Interventions: Drug: Atrovent HFA 42 mcg + Albuterol HFA 200 mcg

INTERVENTIONS:
Drug: Combivent CFC-MDI — 36/206 mcg Four times a day (QID)
  Arms: Combivent CFC-MDI 36/206 microgram-mcg
Drug: Combivent Respimat 20/100 mcg — Open label randomized parallel
  Arms: Combivent Respimat 20/100 microgram(mcg)
Drug: Atrovent HFA 42 mcg + Albuterol HFA 200 mcg — Open label randomized parallel
  Arms: Atrovent HFA 42 mcg + Albuterol HFA

SUMMARY:
The primary objective of this study is to evaluate long-term safety and patient acceptability of COMBIVENT RESPIMAT Inhalation Spray as compared to the COMBIVENT Inhalation Aerosol Chlorofluorocarbon-Metered Dose Inhaler (CFC-MDI) and the free combination of ATROVENT Hydrofluoroalkane (HFA) and albuterol Hydrofluoroalkane (HFA) inhalation aerosols.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization (ICH) Good Clinical Practice (GCP) guidelines prior to participation in the trial.
2. Male or female patients 40 years of age or older.
3. Patients must be current or ex-smokers with a smoking history of 10 pack-years. (Patients who have never smoked cigarettes must be excluded) Pack Years = Number of cigarettes/day x years of smoking 20 cigarettes/pack
4. All patients must have a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) (P95-4381), and must meet the following spirometric criteria at Visit 1:Relatively stable, moderate to severe airway obstruction with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) < 80% of predicted normal and FEV1/Forced Vital Capacity (FVC) < 70%. Spirometry should be done at baseline and approximately 1/2 hour following 4 inhalations of albuterol. Predicted normal values will be calculated according to European Coal and Steel Community (ECSC), European Community for Coal and Steel (ECCS), (R94-1408). For Height measured in inches Males: FEV1 predicted (L) = 4.30 x [height (inches) / 39.37]-0.029 x age (yrs) - 2.49 Females: FEV1 predicted (L) = 3.95 x [height (inches) / 39.37]-0.025 x age (yrs) - 2.60 For Height measured in meters Males: FEV1 predicted (L) = 4.30 x [height (meters)] - 0.029 x age (years) -2.49 Females: FEV1 predicted (L) = 3.95 x [height (meters)] - 0.025 x age (years) - 2.60
5. Patients must be able to perform all study related procedures and maintain study records during the study period as required in the protocol.
6. Patients must be able to inhale medication in a competent manner from the RESPIMAT inhaler and from a metered dose inhaler (MDI).

Exclusion criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with a recent history (i.e., one year or less) of myocardial infarction.
3. Patients who have been hospitalized or being treated for heart failure within the past year.
4. Patients with clinically unstable or life-threatening cardiac arrhythmia requiring intervention or change in drug therapy within the past year.
5. Patients with a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with fully cured squamous cell or treated basal cell carcinoma are allowed).
6. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis.
7. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of a thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1.
8. Patients with a current diagnosis of asthma.
9. Patients with a history of significant alcohol or drug abuse.
10. Patients with known active tuberculosis.
11. Patients using beta blocker medications are excluded. Cardioselective beta blockers are allowed with caution. Beta blocker eye medications for treatment of non-narrow angle glaucoma are allowed.
12. Patients who regularly use daytime oxygen therapy for more than 1 hour per day Continuous Positive Airway Pressure (CPAP for sleep apnea is allowed).
13. Patients using oral corticosteroid medication at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day, except as required for treatment of exacerbation during the study.
14. Pregnant or nursing women.
15. Women of childbearing potential not using a medically approved means of contraception (i.e., oral or injectable contraceptives, intrauterine devices or diaphragm with spermicide, or transdermal hormonal patches). Abstinence will not be accepted as a medically approved means of contraception. Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.
16. Patients with known hypersensitivity to anticholinergic drugs, any other component of the ipratropium bromide/albuterol RESPIMAT solution including Benzalkonium chloride (BAC) and Ethylenediaminetetraacetic acid (EDTA) or the ipratropium bromide/albuterol Chlorofluorocarbons (CFC) MDI or Hydrofluoroalkane (HFA) components.
17. Previous participation in this study. (The patient cannot re-enroll into this study.)
18. Patients who are currently participating in another interventional study.
19. Patients who have taken an investigational drug within 1 month or 6 half lives (whichever is greater) prior to screening.
20. Patients currently in any pulmonary rehabilitation program or scheduled to participate in any such program during the study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (55):
- United States (55):
  - 1012.62.153 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1012.62.145 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1012.62.156 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 1012.62.135 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 1012.62.141 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1012.62.155 Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - 1012.62.126 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1012.62.131 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1012.62.144 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1012.62.123 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1012.62.114 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1012.62.124 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1012.62.139 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1012.62.134 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1012.62.115 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1012.62.146 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1012.62.113 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1012.62.157 Boehringer Ingelheim Investigational Site, Dubuque, Iowa
  - 1012.62.159 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1012.62.116 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1012.62.148 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1012.62.137 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1012.62.132 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1012.62.117 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 1012.62.158 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1012.62.127 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1012.62.129 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1012.62.147 Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - 1012.62.149 Boehringer Ingelheim Investigational Site, Summit, New Jersey
  - 1012.62.112 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1012.62.111 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1012.62.107 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1012.62.120 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1012.62.150 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1012.62.103 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1012.62.104 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1012.62.154 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1012.62.128 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1012.62.130 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1012.62.151 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1012.62.161 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1012.62.109 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1012.62.118 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1012.62.125 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1012.62.140 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1012.62.143 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1012.62.152 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1012.62.102 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1012.62.122 Boehringer Ingelheim Investigational Site, Danville, Virginia
  - 1012.62.119 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1012.62.142 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1012.62.108 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1012.62.133 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1012.62.105 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1012.62.101 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia

REFERENCES:
- [Derived] Ferguson GT, Ghafouri M, Dai L, Dunn LJ. COPD patient satisfaction with ipratropium bromide/albuterol delivered via Respimat: a randomized, controlled study. Int J Chron Obstruct Pulmon Dis. 2013;8:139-50. doi: 10.2147/COPD.S38577. Epub 2013 Mar 19. PMID 23658479

RESULTS

PARTICIPANT FLOW:
Groups:
- Combivent Respimat: ipratropium/albuterol 20/100 micrograms (mcg) 4 per day (qid)
- Combivent Inhalation Aerosol: ipratropium bromide and albuterol sulfate 36/206 mcg qid
- Atrovent + Albuterol Aerosols: ipratropium bromide 34 mcg, albuterol sulfate 180 mcg qid
Period: Overall Study
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Started | 157 (2 pats. in Comb. Inh. Aero. and 3 pats. in Atro+Alb not treated and excluded from the Treated Set) | 156 (2 pats. in Comb. Inh. Aero. and 3 pats. in Atro+Alb not treated and excluded from the Treated Set) | 157 (2 pats. in Comb. Inh. Aero. and 3 pats. in Atro+Alb not treated and excluded from the Treated Set)
Completed | 133 | 118 | 110
Not Completed | 24 | 38 | 47
Not completed — Adverse Event | 12 | 16 | 19
Not completed — Protocol Violation | 2 | 6 | 4
Not completed — Lost to Follow-up | 5 | 3 | 3
Not completed — Withdrawal by Subject | 4 | 6 | 12
Not completed — Not treated | 0 | 2 | 3
Not completed — Other reason (not specified) | 1 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols | Total
Number analyzed (Participants) | 157 | 154 | 154 | 465
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (8.2) | 62.6 (8.9) | 63.0 (9.3) | 62.9 (8.8)
Age, Customized [Number; unit: participants]
  >= 40 to < 65 years | 90 | 91 | 82 | 263
  >= 65 to < 75 years | 51 | 47 | 58 | 156
  >= 75 years | 16 | 16 | 14 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 70 | 57 | 192
  Male | 92 | 84 | 97 | 273
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0 | 0 | 1 | 1
  Black / African American | 9 | 11 | 9 | 29
  White | 148 | 143 | 144 | 435
Height [Mean (Standard Deviation); unit: centimeters] | 170.6 (9.6) | 170.6 (10.4) | 171.1 (10.4) | 170.8 (10.1)
Smoking History [Number; unit: participants]
  Ex-smoker | 83 | 61 | 79 | 223
  Currently smokes | 74 | 93 | 75 | 242
Smoking History (pack years) [Mean (Standard Deviation); unit: pack years] | 53.6 (24.5) | 53.6 (29.7) | 55.6 (25.4) | 54.3 (26.6)
Chronic Obstructive Pulmonary Disease (COPD) Duration [Mean (Standard Deviation); unit: years] | 8.1 (6.7) | 7.3 (6.1) | 7.5 (5.8) | 7.6 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Performance Domain Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 48
Description: Patient acceptability was assessed with the Performance Domain score from the PASAPQ. The score is a mean of 7 items on a scale from 0 (very dissatisfied) to 100 (very satisfied).
Time Frame: 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 134 | 125 | 110
unit on a scale | 87.9 (1.27) | 78.3 (1.31) | 81.7 (1.37)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 9.6, 95% CI [6.02 to 13.19]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 6.2, 95% CI [2.57 to 9.91]

2. Secondary Outcome: Performance Domain Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 3
Description: as for outcome 1
Time Frame: 3 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 152 | 153
unit on a scale | 84.7 (1.07) | 79.4 (1.09) | 77.3 (1.08)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 5.3, 95% CI [2.29 to 8.28]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 7.4, 95% CI [4.41 to 10.39]

3. Secondary Outcome: Performance Domain Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 12
Description: as for outcome 1
Time Frame: 12 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 149 | 149 | 146
unit on a scale | 85.9 (1.14) | 78.0 (1.15) | 76.3 (1.16)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 7.9, 95% CI [4.71 to 11.09]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 9.6, 95% CI [6.44 to 12.83]

4. Secondary Outcome: Performance Domain Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 24
Description: as for outcome 1
Time Frame: 24 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 142 | 142 | 130
unit on a scale | 86.6 (1.15) | 77.5 (1.16) | 78.9 (1.19)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 9.2, 95% CI [5.94 to 12.37]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 7.7, 95% CI [4.44 to 10.96]

5. Secondary Outcome: Performance Domain Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 36
Description: as for outcome 1
Time Frame: 36 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 136 | 132 | 119
unit on a scale | 88.2 (1.22) | 76.9 (1.24) | 80.5 (1.29)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 11.3, 95% CI [7.90 to 14.76]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 7.7, 95% CI [4.23 to 11.23]

6. Secondary Outcome: Overall Satisfaction Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 0
Description: Patient satisfaction was assessed by asking: "Overall, how satisfied are you with your inhaler?". Responses were made on a scale from 1 (very dissatisfied) to 7 (very satisfied).
Time Frame: 0 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 154 | 154
units on a scale | 5.8 (1.21) | 5.9 (1.24) | 5.8 (1.10)

7. Secondary Outcome: Overall Satisfaction Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 3
Description: as for outcome 6
Time Frame: 3 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 152 | 153
unit on a scale | 6.2 (0.08) | 6.1 (0.08) | 5.9 (0.08)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.1167, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.2, 95% CI [-0.05 to 0.42]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.4, 95% CI [0.13 to 0.59]

8. Secondary Outcome: Overall Satisfaction Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 12
Description: as for outcome 6
Time Frame: 12 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 149 | 149 | 146
unit on a scale | 6.2 (0.09) | 6.0 (0.09) | 5.8 (0.09)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.2826, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.1, 95% CI [-0.11 to 0.38]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.4, 95% CI [0.16 to 0.66]

9. Secondary Outcome: Overall Satisfaction Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 24
Description: as for outcome 6
Time Frame: 24 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 142 | 142 | 130
unit on a scale | 6.3 (0.08) | 6.0 (0.08) | 5.8 (0.09)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.4, 95% CI [0.13 to 0.59]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.5, 95% CI [0.25 to 0.71]

10. Secondary Outcome: Overall Satisfaction Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 36
Description: as for outcome 6
Time Frame: 36 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 136 | 132 | 119
unit on a scale | 6.4 (0.08) | 6.0 (0.09) | 5.9 (0.09)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.4, 95% CI [0.18 to 0.65]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.4, 95% CI [0.20 to 0.68]

11. Secondary Outcome: Overall Satisfaction Score From the Patient Satisfaction and Preference Questionnaire (PASAPQ) at Week 48
Description: as for outcome 6
Time Frame: 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 134 | 125 | 110
unit on a scale | 6.3 (0.09) | 6.1 (0.09) | 6.0 (0.09)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.0673, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.2, 95% CI [-0.02 to 0.47]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.0245, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.3, 95% CI [0.04 to 0.54]

12. Secondary Outcome: Clinical COPD Questionnaire (CCQ) Symptom Domain Score at Week 0
Description: CCQ symptom domain score assessed patient feelings or limitations due to their COPD on a scale from 0 (not limited) to 6 (totally limited).
Time Frame: 0 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 153 | 154
units on a scale | 2.8 (1.13) | 2.7 (1.23) | 2.8 (1.13)

13. Secondary Outcome: Clinical COPD Questionnaire (CCQ) Symptom Domain Score at Week 3
Description: as for outcome 12
Time Frame: 3 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 152 | 153
unit on a scale | 2.7 (0.07) | 2.7 (0.07) | 2.8 (0.07)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.5695, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.24 to 0.13]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.3093, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.28 to 0.09]

14. Secondary Outcome: Clinical COPD Questionnaire (CCQ) Symptom Domain Score at Week 12
Description: as for outcome 12
Time Frame: 12 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 150 | 149 | 146
unit on a scale | 2.8 (0.08) | 2.9 (0.08) | 2.8 (0.08)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.3578, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.31 to 0.11]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.7433, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.0, 95% CI [-0.18 to 0.25]

15. Secondary Outcome: Clinical COPD Questionnaire (CCQ) Symptom Domain Score at Week 24
Description: as for outcome 12
Time Frame: 24 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 142 | 142 | 130
unit on a scale | 2.7 (0.08) | 2.8 (0.08) | 2.8 (0.08)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.524, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.29 to 0.15]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.3171, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.34 to 0.11]

16. Secondary Outcome: Clinical COPD Questionnaire (CCQ) Symptom Domain Score at Week 36
Description: as for outcome 12
Time Frame: 36 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 136 | 132 | 119
unit on a scale | 2.7 (0.09) | 2.8 (0.09) | 2.7 (0.09)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.2499, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.38 to 0.10]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.6144, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.31 to 0.18]

17. Secondary Outcome: Clinical COPD Questionnaire (CCQ) Symptom Domain Score at Week 48
Description: as for outcome 12
Time Frame: 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 134 | 125 | 110
unit on a scale | 2.8 (0.09) | 2.7 (0.09) | 2.9 (0.09)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.5142, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.1, 95% CI [-0.16 to 0.33]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.2691, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.39 to 0.11]

18. Secondary Outcome: Physician's Global Evaluation at Week 0
Description: Physicians evaluated the patient's overall clinical condition on a scale ranging from "poor" (score 1 or 2) to "excellent" (score 7 or 8).
Time Frame: 0 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 154 | 154
units on a scale | 5.1 (1.18) | 4.9 (1.22) | 4.9 (1.26)

19. Secondary Outcome: Physician's Global Evaluation at Week 3
Description: as for outcome 18
Time Frame: 3 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 152 | 152
unit on a scale | 5.0 (0.07) | 5.1 (0.07) | 5.1 (0.07)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.6236, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.0, 95% CI [-0.23 to 0.14]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.3342, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.28 to 0.09]

20. Secondary Outcome: Physician's Global Evaluation at Week 12
Description: as for outcome 18
Time Frame: 12 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 150 | 148 | 146
unit on a scale | 5.1 (0.08) | 5.2 (0.08) | 5.0 (0.08)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.1884, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.36 to 0.07]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.6978, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.0, 95% CI [-0.17 to 0.26]

21. Secondary Outcome: Physician's Global Evaluation at Week 24
Description: as for outcome 18
Time Frame: 24 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 142 | 142 | 130
unit on a scale | 5.1 (0.08) | 5.2 (0.08) | 5.2 (0.08)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.4197, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.32 to 0.13]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.3949, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.33 to 0.13]

22. Secondary Outcome: Physician's Global Evaluation at Week 36
Description: as for outcome 18
Time Frame: 36 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 136 | 132 | 118
unit on a scale | 5.1 (0.09) | 5.2 (0.09) | 5.2 (0.09)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.299, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.38 to 0.12]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.1404, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.2, 95% CI [-0.44 to 0.06]

23. Secondary Outcome: Physician's Global Evaluation at Week 48
Description: as for outcome 18
Time Frame: 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 133 | 125 | 108
unit on a scale | 5.2 (0.09) | 5.3 (0.09) | 5.1 (0.10)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.463, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.36 to 0.16]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.3824, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.1, 95% CI [-0.15 to 0.38]

24. Secondary Outcome: Change From Baseline in FEV1 at Day 1
Description: Change from test-day baseline in Forced Expiratory Volume in 1 second (FEV1) at 1 hour post dose on test day 1.
Time Frame: baseline, day 1
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 154 | 154
liters | 0.22 (0.015) | 0.21 (0.015) | 0.21 (0.015)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.8282, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.0, 95% CI [-0.036 to 0.045]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.6587, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.01, 95% CI [-0.032 to 0.050]

25. Secondary Outcome: Change From Baseline in FEV1 at Week 12
Description: Change from test-day baseline in Forced Expiratory Volume in 1 second (FEV1) at 1 hour post dose at Week 12
Time Frame: baseline, 12 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 145 | 144 | 136
liters | 0.23 (0.016) | 0.19 (0.016) | 0.20 (0.017)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.1185, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.04, 95% CI [-0.009 to 0.081]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.2651, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.03, 95% CI [-0.020 to 0.072]

26. Secondary Outcome: Change From Baseline in FEV1 at Week 24
Description: Change from test-day baseline in Forced Expiratory Volume in 1 second (FEV1) at 1 hour post dose at Week 24
Time Frame: baseline, 24 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 138 | 134 | 124
liters | 0.20 (0.016) | 0.21 (0.016) | 0.21 (0.017)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.5852, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.01, 95% CI [-0.058 to 0.033]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.7242, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.01, 95% CI [-0.054 to 0.038]

27. Secondary Outcome: Change From Baseline in FEV1 at Week 48
Description: Change from test-day baseline in Forced Expiratory Volume in 1 second (FEV1) at 1 hour post dose at Week 48
Time Frame: baseline, 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 133 | 121 | 108
liters | 0.22 (0.019) | 0.16 (0.019) | 0.23 (0.020)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.0328, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.06, 95% CI [0.005 to 0.110]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.8896, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.00, 95% CI [-0.058 to 0.050]

28. Secondary Outcome: Change From Baseline in FVC at Day 1
Description: Change from test-day baseline in Forced Vital Capacity (FVC) at 1 hour post dose on test day 1.
Time Frame: baseline, day 1
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 154 | 154
liters | 0.37 (0.026) | 0.34 (0.027) | 0.36 (0.027)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.402, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.03, 95% CI [-0.042 to 0.105]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.659, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.02, 95% CI [-0.057 to 0.090]

29. Secondary Outcome: Change From Baseline in FVC at Week 12
Description: Change from test-day baseline in Forced Vital Capacity (FVC) at 1 hour post dose at Week 12
Time Frame: baseline, 12 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 145 | 144 | 136
liters | 0.38 (0.027) | 0.31 (0.027) | 0.35 (0.027)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.0893, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.06, 95% CI [-0.010 to 0.139]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.5424, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.02, 95% CI [-0.052 to 0.099]

30. Secondary Outcome: Change From Baseline in FVC at Week 24
Description: Change from test-day baseline in Forced Vital Capacity (FVC) at 1 hour post dose at Week 24
Time Frame: baseline, 24 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 138 | 134 | 124
liters | 0.33 (0.030) | 0.35 (0.030) | 0.35 (0.031)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.6396, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.02, 95% CI [-0.104 to 0.064]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.6455, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.02, 95% CI [-0.106 to 0.066]

31. Secondary Outcome: Change From Baseline in FVC at Week 48
Description: Change from test-day baseline in Forced Vital Capacity (FVC) at 1 hour post dose at Week 48
Time Frame: baseline, 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 133 | 121 | 108
liters | 0.35 (0.032) | 0.30 (0.033) | 0.37 (0.034)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.2596, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.05, 95% CI [-0.038 to 0.141]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.6659, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.02, 95% CI [-0.112 to 0.071]

32. Secondary Outcome: Mean Number of Puffs of Daily Rescue Medication Use in Two Weeks Prior to Week 0
Description: Mean number of puffs of daily rescue medication use (albuterol use per 24 hour period) in two weeks prior to week 0
Time Frame: 0 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Mean (Standard Deviation); unit: number of puffs
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 153 | 154
number of puffs | 2.1 (2.63) | 1.5 (2.23) | 1.9 (2.70)

33. Secondary Outcome: Mean Number of Puffs of Daily Rescue Medication Use in Two Weeks Prior to Week 3
Description: Mean number of puffs of daily rescue medication use (albuterol use per 24 hour period) in two weeks prior to week 3
Time Frame: 3 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 151 | 152
number of puffs | 1.7 (0.10) | 1.8 (0.11) | 1.7 (0.11)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.476, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.40 to 0.19]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.6976, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.35 to 0.23]

34. Secondary Outcome: Mean Number of Puffs of Daily Rescue Medication Use in Two Weeks Prior to Week 12
Description: Mean number of puffs of daily rescue medication use (albuterol use per 24 hour period) in two weeks prior to week 12
Time Frame: 12 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 147 | 149 | 145
number of puffs | 1.9 (0.14) | 1.9 (0.14) | 1.7 (0.14)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.9506, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.0, 95% CI [-0.40 to 0.37]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.2362, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.2, 95% CI [-0.15 to 0.62]

35. Secondary Outcome: Mean Number of Puffs of Daily Rescue Medication Use in Two Weeks Prior to Week 24
Description: Mean number of puffs of daily rescue medication use (albuterol use per 24 hour period) in two weeks prior to week 24
Time Frame: 24 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 142 | 143 | 129
number of puffs | 2.1 (0.15) | 2.0 (0.15) | 1.6 (0.16)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.5645, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.1, 95% CI [-0.30 to 0.54]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.0163, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.5, 95% CI [0.10 to 0.95]

36. Secondary Outcome: Mean Number of Puffs of Daily Rescue Medication Use in Two Weeks Prior to Week 36
Description: Mean number of puffs of daily rescue medication use (albuterol use per 24 hour period) in two weeks prior to week 36
Time Frame: 36 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 136 | 131 | 116
number of puffs | 1.9 (0.15) | 2.1 (0.15) | 1.8 (0.16)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.4339, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.2, 95% CI [-0.60 to 0.26]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.4886, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.2, 95% CI [-0.28 to 0.59]

37. Secondary Outcome: Mean Number of Puffs of Daily Rescue Medication Use in Two Weeks Prior to Week 48
Description: Mean number of puffs of daily rescue medication use (albuterol use per 24 hour period) in two weeks prior to week 48
Time Frame: 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 133 | 122 | 110
number of puffs | 2.0 (0.16) | 2.1 (0.16) | 1.8 (0.16)
Statistical Analysis 1: Comparison: Combivent Respimat vs Combivent Inhalation Aerosol; Comparison of Combivent Respimat versus Combivent Inhalation Aerosol; Test type: Superiority or Other; p = 0.7637, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = -0.1, 95% CI [-0.50 to 0.37]
Statistical Analysis 2: Comparison: Combivent Respimat vs Atrovent + Albuterol Aerosols; Comparison of Combivent Respimat versus Atrovent + Albuterol Aerosols; Test type: Superiority or Other; p = 0.3755, Mixed Models Analysis; Adjusted for baseline and baseline-by-test-day interaction; Mean Difference (Final Values) = 0.2, 95% CI [-0.24 to 0.65]

38. Secondary Outcome: Number of Patients Having Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Time Frame: 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Number; unit: participants
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 154 | 154
participants
  None | 118 (118) | 113 (113) | 110 (110)
  1 exacerbation | 27 | 32 | 37
  2 exacerbations | 7 | 9 | 5
  3 exacerbations | 3 | 0 | 2
  4 exacerbations | 1 | 0 | 0
  5 or more exacerbations | 1 | 0 | 0

39. Secondary Outcome: Number of Patients Having Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Leading to Hospitalization
Time Frame: 48 weeks
Population: Treated Set is defined as all patients who were randomized and received study drug
Measure: Number; unit: participants
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Number analyzed (Participants) | 157 | 154 | 154
participants
  None | 147 (147) | 148 (148) | 146 (146)
  1 exacerbation | 9 | 6 | 8
  2 exacerbations | 0 | 0 | 0
  3 or more exacerbations | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first drug intake until one day after last drug intake
Arm/Group | Combivent Respimat | Combivent Inhalation Aerosol | Atrovent + Albuterol Aerosols
Serious Adverse Events (participants affected / at risk) | 23/157 | 20/154 | 25/154
Other Adverse Events (participants affected / at risk) | 68/157 | 76/154 | 71/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combivent Respimat (N=157) | Combivent Inhalation Aerosol (N=154) | Atrovent + Albuterol Aerosols (N=154)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Pituitary haemorrhage (Endocrine disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 2
Appendicitis perforated (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac enzymes increased (Investigations) | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combivent Respimat (N=157) | Combivent Inhalation Aerosol (N=154) | Atrovent + Albuterol Aerosols (N=154)
Bronchitis (Infections and infestations) | 11 | 10 | 9
Nasopharyngitis (Infections and infestations) | 6 | 8 | 9
Sinusitis (Infections and infestations) | 6 | 10 | 11
Upper respiratory tract infection (Infections and infestations) | 16 | 19 | 14
Insomnia (Psychiatric disorders) | 2 | 8 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 23 | 26 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.